CLINICAL TRIAL: NCT02350556
Title: Interest of Evaluating the Movement of the Center of Mass in a Dynamic Avoidance Task as the Endpoint of the Dynamic Equilibrium of Hemiplegic Patients
Acronym: EQHEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-A00097-40
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hemiplegic Patients
MeSH Terms: interventions — Physical Therapy Modalities

ARMS (2):
- hemiplegic patients (Other): Dynamic Avoidance Task
  Interventions: Other: Dynamic Avoidance Task; Procedure: physical therapy; Device: 3D motion on optoelectronic device
- healthy volunteers (Other): Dynamic Avoidance Task
  Interventions: Other: Dynamic Avoidance Task; Procedure: physical therapy; Device: 3D motion on optoelectronic device

INTERVENTIONS:
Other: Dynamic Avoidance Task
Procedure: physical therapy
Device: 3D motion on optoelectronic device

SUMMARY:
For several years, the postural disorders assessment in hemiplegic patients was conducted through force plate, using the center of plantar pressure displacement in a static position.

These are widely used in physical therapy both for assessment and rehabilitation of patients with balance disorders.

For hemiplegic patients, an asymmetric distribution support on each foot and an increased surface area of postural sways (more marked on the medio lateral axis) are observed.

These studies, based on the study of plantar pressure ,are not enough to providea full description of the spatio-temporal organization of postural components in hemiplegic patients.

Indeed, postural stabilometric evaluation is based on a simplification of the human skeleton by considering it as a simple inverted pendulum swinging on his ankles.

This simplified model can't be used in dynamic assessment because of the simultaneous contributions of several joints during movement. This restricts its clinical interest because patients are more exposed to imbalances and falls in dynamic situations. Thus, the hip angular movement results in a center plantar pressure displacementwhich is impossible to discriminate from the ankle axis movement using stabilometric signal only.

Thus, it seemed interesting to study another variable valid in dynamic conditions : the displacement of center of mass during a dynamic balancing task. This variable is obtained through 3D motion capture of the different segments of the human body. The dynamic test is a dynamic postural assessment following ball avoidance from three different directions. The center of mass displacement will be compared with a functional test known to be representative of dynamic balance of the individual capacities: The Timed Up and Go test (TUG).

All of this data aims to improve the hemiplegic postural assessment for physical therapy and to help develop new rehabilitative approaches.

ELIGIBILITY:
Inclusion Criteria:

-

For hemiplegic patients:

* Aged between 18-80 years of age, men and women
* Left or right hemispheric sustentoriel stroke :

oIschemic or hemorragic oFirst symptomatic episode or TIA without consequences oBetween one month and one year since the stroke

* Balance standing > 30 sec without assistance in closed eyes condition
* FAC score included between 3 and 7
* Triceps Spasticity strictly less than 3 on the Modified Ashworth Scale with heel on the ground and an adductor spasticity up to 3 on the same scale.
* Free, informed and written consent signed by the investigator and by the patient or one of his/her relatives (in the case of a patient able to understand the information and to express his/her consent but with motor difficulties resulting in the inability to sign)

For healthy volunteers :

* Aged between 18-85 years of age, men or women, age-matched ( +/- 5 years ) with stroke patients
* Without a balance disorder
* Affiliated to social security
* Free, informed and written consent

Exclusion Criteria:

For hemiplegic patients:

* History of event affecting postural balance (orthopedic, rheumatological, neurological, ENT ...) before the stroke
* Pregnant women
* Patient with tiredness incompatible with the tests and instrumental assessments
* Patients under legal protection (according to French law) and detainees.
* Patients physically or mentally unable of giving informed consent

For healthy volunteers :

* History of event affecting postural balance (orthopedic, rheumatological, neurological, ENT ...)
* Receiving a psychotropic treatment (antidepressant, antipsychotic, anxiolytic)
* Pregnant women
* Within the period of exclusion in the French national register of persons suitable for biomedical research
* Patients under legal protection (according to French law) and detainees.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the lateral displacement of the center of mass (CoM) in the frontal plane, obtained after recording the 3D motion using an optoelectronic device | dynamic avoidance test in 7 days

SECONDARY OUTCOMES:
- to the functional level and the balance obtained from the test: Timed Up and Go test (TUG). This comparison will be made regarding the completion time of the test and the functional score in the Get Up and Go test. | inclusion (0)
- using dynamic assessments : Maximum front displacement of the Plantar pressure center (CP) resultant when avoiding the central ball, | dynamic avoidance test in 7 days
- Using static assessments : Postural asymmetry obtained by calculating the percentage of body weight distribution on each leg during the static postural initial assessment on force plate | Inclusion (0)
The ABS TUG score (being validated) will also be compared to the lateral displacement of the center of mass (CoM). | inclusio (0)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes Pontchaillou, Rennes, France